CLINICAL TRIAL: NCT03502772
Title: The Effects of Clinical Pilates Training on Walking, Balance, Fall Risk, Respiratory and Cognitive Functions in Persons With Multiple Sclerosis: A Randomized Controlled Trial
Brief Title: Clinical Pilates Training for Persons With Multiple Sclerosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dokuz Eylul University (Other)
Collaborators: Izmir Katip Celebi University (Other)
Responsible Party: Principal Investigator, Turhan Kahraman, Principal Investigator, Dokuz Eylul University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3183-GOA
Record Dates: First submitted 2018-04-11; First posted 2018-04-19 (Actual); Last update posted 2018-04-19 (Actual); Status verified 2018-04

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis | interventions — Exercise Movement Techniques

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pilates exercises group (Experimental)
  Interventions: Other: Pilates exercises
- Home exercise program group (Active Comparator)
  Interventions: Other: Home exercise program

INTERVENTIONS:
Other: Pilates exercises — Clinical Pilates training program will be given one session in a week for 8 weeks plus two days home exercise program. Group exercise sessions will be performed. The sessions will be supervised by a physiotherapist who is certified.
  Arms: Pilates exercises group
Other: Home exercise program — written exercises that matched the aims of the Pilates exercises, 3 times per week for 8 weeks. These exercises reflect routine clinical practice (flexibility, strength, and balance exercises).
  Arms: Home exercise program group

SUMMARY:
Multiple sclerosis (MS) is a chronic-progressive and neurodegenerative disease. Thus, exercise programs are needed to maintain and increase functional status of persons with MS (pwMS). Pilates exercises designed by physiotherapist can enhance participation and functionality in pwMS. The aim is to investigate the effects of a clinical Pilates training on balance, walking, fall risk, respiratory and cognitive functions in pwMS.

Forty-two pwMS will be included in this randomized controlled trial. Participants will be divided into two groups with stratified randomization. Pilates exercises group (n=21) will receive therapy once a week for 8 weeks plus home exercise programme. The home exercise program group (n = 21) will be given written exercises that matched the aims of the Pilates exercises and the program compliance will be monitored by telephone calls once a week. The assessments will be done twice at the beginning and at the end of the treatment. The outcome measures include the Timed 25-Foot Walk (T25FW), Six-Minute Walk Test (6MWT), Timed Up and Go (TUG), TUG cognitive and manual forms, 12-Item Multiple Sclerosis Walking Scale (MSWS-12), Curl-Up Test (CUT), Falls Efficacy Scale-International (FES-I), Activities-specific Balance Confidence (ABC) Scale, respiratory muscle strength assessment, Brief International Cognitive Assessment for MS (BICAMS).

ELIGIBILITY:
Inclusion Criteria:

* a diagnosis of definite MS
* an age over than 18 years
* walking independently 100 meters
* willingness to participate in the study

Exclusion Criteria:

* any neurological disease other than multiple sclerosis
* relapse within 3 months
* having orthopaedic disorders that could negatively affect gait and balance
* having cardiopulmonary disorders
* diagnosed cognitive and psychiatric problems
* current and recent (within the last 6 months) participation in a core stability based exercise program

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2017-04-03 (Actual); Primary Completion 2017-12-29 (Actual); Study Completion 2017-12-29 (Actual)

PRIMARY OUTCOMES:
12-Item MS Walking Scale | Change from Baseline at 8 weeks
  The 12-item Multiple Sclerosis Walking Scale (MSWS-12) is a self-report measure of the impact of multiple sclerosis on the individual's walking ability. The first 3 items are scored 1 - 3, and the other 9 items are scored 1 - 5. Scores on the 12 items are summed. The minimum score is 12 and the maximum score is 54. Higher the score, greater the impacted walking quality.

SECONDARY OUTCOMES:
Six-Minute Walk Test | Change from Baseline at 8 weeks
Timed 25-Foot Walk | Change from Baseline at 8 weeks
Timed-Up and Go | Change from Baseline at 8 weeks
Limits of Stability Test | Change from Baseline at 8 weeks
Postural Stability Test | Change from Baseline at 8 weeks
Fall Risk Index | Change from Baseline at 8 weeks
Falls Efficacy Scale-International | Change from Baseline at 8 weeks
  Falls Efficacy Scale-International is a 16-item self-administered questionnaire designed to assess fear of falling. Items are scored a 1 if they are not at all concerned about falling going up to 4 if they are very concerned during each activity: 1 = Not at all concerned, 2 = Somewhat concerned, 3 = Fairly concerned, 4 = Very concerned. Item scores are summed to calculate a range of total score from minimum 16 to maximum 64. Higher the score, greater the fear of falling.
Activities-Specific Balance Confidence Scale | Change from Baseline at 8 weeks
  The Activities-Specific Balance Confidence Scale is a subjective measure of confidence in performing various ambulatory activities without falling or experiencing a sense of unsteadiness. 16-item self-report measure in which patients rate their balance confidence for performing activities. This stem is used to lead into each activity considered: "How confident are you that you will not lose your balance or become unsteady when you..." Items are rated on a rating scale that ranges from 0 - 100. Score of zero represents no confidence, a score of 100 represents complete confidence. Overall score is calculated by adding item scores and then dividing by the total number of items.
Curl-up Test | Change from Baseline at 8 weeks
Maximum Inspiratory Pressure | Change from Baseline at 8 weeks
Maximum Expiratory Pressure | Change from Baseline at 8 weeks
Symbol Digit Modalities Test | Change from Baseline at 8 weeks
California Verbal Learning Test-II | Change from Baseline at 8 weeks
Brief Visuospatial Memory Test Revised | Change from Baseline at 8 weeks
Expanded Disability Status Scale | At Baseline
  The Expanded Disability Status Scale is a method of quantifying disability in multiple sclerosis and monitoring changes in the level of disability over time. It is widely used in clinical trials and in the assessment of people with multiple sclerosis. The Expanded Disability Status Scale ranges from 0 to 10 in 0.5 unit increments that represent higher levels of disability. Scoring is based on an examination by a neurologist. Expanded Disability Status Scale steps 1.0 to 4.5 refer to people with multiple sclerosis who are able to walk without any aid. Expanded Disability Status Scale steps 5.0 to 9.5 are defined by the impairment to walking. Persons with multiple sclerosis with Expanded Disability Status Scale steps 6 and below will be participated in the study.

CONTACTS AND LOCATIONS:
Locations (1):
- Dokuz Eylul University Hospital, MS Outpatient Clinic, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided